CLINICAL TRIAL: NCT05113654
Title: Sleep Disorders in Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: WI_SleepIPF_169/2015
Record Dates: First submitted 2021-10-04; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IPF: Patients with idiopathic pulmonary fibrosis
  Interventions: Diagnostic Test: Sleep study
- COPD: Patients with chronic obstructive pulmonary disease
  Interventions: Diagnostic Test: Sleep study
- Healthy: Healthy controls
  Interventions: Diagnostic Test: Sleep study

INTERVENTIONS:
Diagnostic Test: Sleep study — Nocturnal polysomnography or polygraphy to assess sleep-related breathing disorder and other sleep disorders

SUMMARY:
This diagnostic observational study was conducted to (1) investigate the prevalence of sleep-related breathing disorders and other sleep disorders in idiopathic pulmonary fibrosis in comparison to COPD, (2) identify characteristics of symptomatic and prognostic significance in idiopathic pulmonary fibrosis with/without sleep disorders, and (3) evaluate different tools for their ability to assess the risk of co-existing sleep disorders in idiopathic pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* written informed consent
* IPF cohort: Documented history of IPF with definite or possible UIP pattern and signs of emphysema below 10% by HRCT (IPF diagnosis according to 2011 ATS/ERS IPF guidelines)
* COPD cohort: Documented history of COPD Stage II Group A or B, Stage III or IV, Group C or D (GOLD 2014)

Exclusion Criteria:

* Long-term oxygen therapy
* Heart failure NYHA stages III and IV
* Left ventricular ejection fraction ≤ 45%
* Pregnancy and/or lactation
* Acute and/or life-threatening illness (instable angina pectoris, acute pulmonary arterial embolism, myocardial infarction, malignant tumor requiring treatment)
* Current drug or alcohol abuse
* Any medical, psychological or other condition impairing the patient's ability to provide informed consent
* IPF cohort: Acute exacerbation of IPF
* IPF cohort: Concomitant lung/airway diseases other than IPF (signs of emphysema >10% by HRCT)
* COPD cohort: Acute exacerbation of COPD
* COPD cohort: Concomitant lung/airway diseases other than COPD (e.g. Asthma bronchiale)
* Healthy cohort: Documented history of structural airway or lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants were recruited from clinical routine patients.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with any kind of sleep disorder according to the International Classification of Sleep Disorders (ICSD-3) | For individual assessment of sleep disorders: one night (between 5 and 9 hours), for overall number of patients: entire study duration (37 months)
  Sleep disorders defined by the International Classfication of Sleep Disorders are diagnosed by a single sleep study (polysomnography or polygraphy), lasting between 5 and 9 hours for each individual participant. The number of patients for whom at least one sleep disorder is diagnosed, is used to calculate the prevalence of sleep disorders among each patient group.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Randerath, Prof. Dr., Principal Investigator — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- Wissenschaftliches Institut Bethanien e.V., Solingen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No